CLINICAL TRIAL: NCT03117933
Title: Randomised Phase II Trial of Olaparib, Chemotherapy or Olaparib and Cediranib in Patients With Platinum-resistant Ovarian Cancer
Brief Title: Olaparib +/- Cediranib or Chemotherapy in Patients With Platinum-resistant Ovarian Cancer
Acronym: OCTOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_062; 2016-000559-28 (EudraCT Number); 16/LO/2150 (Other: Research Ethics Committee)
Record Dates: First submitted 2017-03-21; First posted 2017-04-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer
Keywords: BRCA1/2 mutation; Platinum resistance
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; cediranib; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Randomised open label trial with 3 arms, stratified for prior PARP use, prior anti-angiogenic use and BRCA status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: Paclitaxel (Active Comparator): Paclitaxel, IV weekly, 80mg/m2; until progression
  Interventions: Drug: Paclitaxel
- B: Olaparib (Experimental): Olaparib, oral, 300mg twice daily; until progression
  Interventions: Drug: Olaparib
- C: Olaparib and Cediranib (Experimental): Olaparib, oral, 300mg twice daily and Cediranib, tablet, 20mg once daily; until progression
  Interventions: Drug: Olaparib; Drug: Cediranib

INTERVENTIONS:
Drug: Olaparib — Tablet, 100mg and 150mg
  Arms: B: Olaparib; C: Olaparib and Cediranib
Drug: Cediranib — Tablet 15mg and 20mg
  Arms: C: Olaparib and Cediranib
Drug: Paclitaxel — Intravenous (IV)
  Arms: A: Paclitaxel

SUMMARY:
The trial will compare the drugs olaparib and cediranib with standard chemotherapy in platinum resistant ovarian cancer. Patients will be randomised to one of three treatment groups: olaparib only, olaparib and cediranib and the control group paclitaxel. The aim is to compare efficacy of the 3 treatments and also how well each treatment is tolerated including the participants quality of life.

DETAILED DESCRIPTION:
Olaparib is a PARP inhibitor which targets BRCA1/2 mutated tumour cells and cediranib is an anti-angiogenic drug which reduces blood supply to the tumour, suppressing tumour viability. Phase I/II trials of both drugs have shown these are well tolerated alone or in combination in ovarian cancer.

The trial aims to compare the efficacy of the combination and of olaparib alone with paclitaxel chemotherapy and whether the olaparib/cediranib combination is better tolerated thus improving quality of life. Secondly standard paclitaxel chemotherapy must be administered weekly at hospital whereas the olaparib/cediranib combination can be administered at home potentially also improving patient quality of life.

Participants' tumours will be resistant to platinum based therapies. Participants will be randomised into one of the 3 treatment arms after stratification for prior PARP/anti-angiogenic treatments/BRCA status. Participants will be on trial up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, age ≥ 16 years with relapsed epithelial ovarian, primary peritoneal or fallopian tube cancer who have relapsed within 12 months of previous platinum-based therapy. Their most recent chemotherapy does not have to have been platinum-based.
2. Patients can have received prior PARP inhibitor, but there must be a > 6 month interval since treatment.
3. Patients can have received prior antiangiogenic therapy, but there must be a > 6 month interval since treatment; except for bevacizumab where a 6 week interval is required.
4. Measurable disease by RECIST Version 1.1 performed in past 4 weeks. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
5. Sufficient archival tissue confirming histological diagnosis available.
6. ECOG PS 0-2
7. Able to swallow and retain oral medications.
8. Life expectancy > 12 weeks in terms of disease related mortality
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. Written (signed and dated) informed consent prior to any study specific procedures and be capable of co-operating with protocol.
11. Patients must have

    • Haemoglobin ≥ 9.0 g/dL and no blood transfusions in the 28 days prior to randomisation
12. Patients must have normal organ and bone marrow function measured within 14 days prior to administration of study treatment as defined below:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count > 100 x 109/L
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
    * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) or calculated creatinine clearance >50 ml/min calculated using Cockroft-Gault, Jelliffe or Wright (see Appendix 4)
    * Urine dipstick for proteinuria <2+. If urine dipstick is ≥ 2+ on two occasions more than one week apart then a 24-hour urine must demonstrate ≤ 1 g of protein in 24 hours or protein/creatinine ratio < 1.5.

Exclusion Criteria:

1. Received previous single agent weekly paclitaxel for relapsed disease.
2. Pregnant or breast-feeding women or women of childbearing potential unless effective methods of contraception are used during the trial and for 6 months after stopping treatment. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Pregnancy test will be performed monthly in women of child bearing potential.

   Postmenopausal is defined as:
   * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
   * LH and FSH levels in the post-menopausal range for women under 50,
   * radiation-induced oophorectomy with last menses >1 year ago,
   * chemotherapy-induced menopause with >1 year interval since last menses, or surgical sterilisation (bilateral oophorectomy or hysterectomy).
3. Treatment with any other investigational agent, systemic chemotherapy, or participation in another interventional clinical trial within 28 days prior to enrolment.
4. Radiotherapy within 2 weeks from the last dose prior to study treatment
5. Started a stable dose of bisphosphonates for bone metastases less than 4 weeks prior to treatment with study drug e.g. patient is eligible and can continue to take bisphosphonates if these were started at least 4 weeks prior to treatment with study drug.
6. Concomitant use of known CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.
7. Concomitant use of potent inducers of CYP3A4 such as rifampicin, carbamazepine, phenobarbital, phenytoin and St. John Wort.
8. Persistent toxicities (>=CTCAE grade 2) caused by previous cancer therapy with the exception of alopecia.
9. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
10. Blood transfusions within 1 month prior to study start
11. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
12. Patients with symptomatic, untreated, uncontrolled brain or meningeal metastases or tumour.

    a. A scan to confirm the absence of brain metastases is not required. b. Patients with radiological evidence of stable brain metastases are eligible, providing that they are asymptomatic and: i. Do not require corticosteroids, or ii. Have previously been treated with corticosteroids, with clinical and radiological evidence of stabilisation at least 10 days after discontinuation of steroids iii. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment.
13. Major surgery within 14 days of starting study treatment
14. Patients who have not recovered from any effects of any major surgery.
15. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan
16. Any psychiatric disorder that prohibits obtaining informed consent.
17. Left Ventricular Ejection Fraction (LVEF) < institutional lower limit of normal, when:

    i. Prior treatment with anthracyclines (excluding liposomal doxorubicin) ii. Prior treatment with trastuzumab iii. A NYHA classification of II controlled with treatment (see Appendix 2) iv. Prior central thoracic RT, including RT to the heart v. History of myocardial infarction within the prior 12 months
18. Poorly controlled hypertension (persistently elevated > 150/100mmHg, either systolic or diastolic or both, despite anti-hypertensive medication)
19. History of inflammatory bowel disease
20. History of cerebrovascular accident (including transient ischaemic attacks) within last 12 months.
21. Gastro intestinal impairment that could affect ability to take, or absorption of, oral medicines including sub- acute or complete bowel obstruction
22. Evidence of severe or uncontrolled cardiac disease
23. Evidence of active bleeding or bleeding diathesis. Defined as significant haemorrhage (>30mL bleeding/episode in previous 3 months) or haemoptysis (>5mL fresh blood in previous 4 weeks)
24. Known treatment-limiting hypersensitivity to cediranib, olaparib, paclitaxel or any of its excipients
25. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
26. Any other active malignancy, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions, requiring treatment/or whose prognosis will prevent readout from trial endpoints.
27. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.

28 Immunocompromised patients e.g., patients who are taking immunosuppressive drugs.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | up to 18 months
  Progression free survival (PFS), measured as time from date of randomisation to RECIST-defined progression or death from any cause (whichever is first)

SECONDARY OUTCOMES:
Adverse events | up to 18 months
  Adverse events using CTCAE v4.03
Overall Survival | 12 & 18 months
  Overall Survival
Objective Response Rate | up to 18 months
  Objective Response Rate based on RECIST v1.1
Objective Response Rate | up to 18 months
  Objective Response Rate based GCIG CA125
Quality of Life Outcomes | up to 18 months
  Quality of Life Outcomes based on EORTC-QLQ C30
Quality of Life Outcomes | up to 18 months
  Quality of Life Outcomes based on EQ5D
Quality of Life Outcomes | up to 18 months
  Quality of Life Outcomes based on OV28.

CONTACTS AND LOCATIONS:
Locations (14):
- United Kingdom (14):
  - Belfast City Hospital, Belfast, County Antrim
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - City Hospital Nottingham, Nottingham, Nottinghamshire
  - Royal Surrey County Hospital, Guildford, Surrey
  - Royal United Hospital, Bath
  - Velindre, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Clatterbridge Cancer Centre, Liverpool
  - St Bartholomew's, London
  - Hammersmith Hospital, London
  - Royal Marsden Chelsea & Sutton, London
  - University College London, London
  - The Christie, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Mansouri A, McGregor N, Dunn R, Dobbie S, Holmes J, Collins L, Nicum S. Randomised phase II trial of olaparib, chemotherapy or olaparib and cediranib in patients with platinum-resistant ovarian cancer (OCTOVA): a study protocol. BMJ Open. 2021 Jan 15;11(1):e041463. doi: 10.1136/bmjopen-2020-041463. PMID 33452192